CLINICAL TRIAL: NCT03838302
Title: Evaluation of Female Sexual Functions With Validated Measurement Scale (Female Sexual Function Index) After Transvaginal Versus Trocars Extraction of Tissue by Laparoscopic Surgery With Uterus Preservation
Brief Title: Evaluation of Sexual Functions With Validated Measurement Scale After Transvaginal Extraction of Tissue by Laparoscopic Surgery With Uterus Preservation (FSF-TVE)
Acronym: FSF-TVE
Status: Not yet recruiting | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: FSF-TVE
Record Dates: First submitted 2019-02-09; First posted 2019-02-12 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Transvaginal Tissue Extraction
Keywords: Sexual functioning; Laparoscopy; Colpotomy; Specimen retrieval; Transvaginal extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transvaginal retrieval: Transvaginal retrieval via a posterior colpotomy for removing tissue by laparoscopic surgery with uterus preservation
  Interventions: Procedure: Transvaginal tissue retrieval via a posterior colpotomy
- Transabdominal retrieval: Transabdominal retrieval via trocar for removing tissue by laparoscopic surgery with uterus preservation
  Interventions: Procedure: Transabdominal retrieval via trocar

INTERVENTIONS:
Procedure: Transvaginal tissue retrieval via a posterior colpotomy — Transvaginal retrieval via a posterior colpotomy for removing tissue by laparoscopic surgery with uterus preservation
  Groups: Transvaginal retrieval
Procedure: Transabdominal retrieval via trocar — Transabdominal retrieval via trocar for removing tissue by laparoscopic surgery with uterus preservation
  Groups: Transabdominal retrieval

SUMMARY:
The retrieval of tissues removed by laparoscopic surgery larger than trocars caliber, with preservation of the uterus, required for a long time intraperitoneal electromechanical morcellation, until the Food and Drug Administration expressed concern about intraperitoneal dissemination of malignant cells, in the case of unrecognized sarcomas.

Transvaginal contained tissue extraction via a posterior colpotomy and manual morcellation in the bag is one of the possible alternatives.

Available data suggested the effectiveness and safety of this technique, also in terms of time and costs, without a increased risk intra and post-operative complications.

The available evidence shows the lack of sequelae also on fertility and sexual function.

Nevertheless, sexual function has never been evaluated qualitatively in all its aspects nor quantitatively with a validated measurement scale, which can allow us to inform the consequences on the real risk of implications on sexual function determined by vaginal incision. In view of these elements, the aim of the investigator's study is to compare patients in whom laparoscopic tissue removal has been carried out with posterior colpotomy or without it with removal from the trocars.

ELIGIBILITY:
Inclusion Criteria:

* Benign uterine and adnexal pathology
* Preservation of the uterus
* Sexually active women
* Premenopausal women

Exclusion Criteria:

* Pelvic inflammatory disease, endometriosis and pre-existing dyspareunia or chronic pelvic pain of any origin
* Previous Hysterectomy
* Other gynecological and non-gynecological (chronic endocrine, metabolic, autoimmune, neoplastic diseases, psychopathology, mental and sensory-motor disabilities) comorbidities
* Language barrier

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing laparoscopic management for myomas or adnexal disease and with specimen retrieval by transvaginal extraction or transbdominal extraction through trocar.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | Change from baseline (before surgery) and 2 months after surgery
  The Female Sexual Function Index (FSFI) is a brief questionnaire measure of sexual functioning in women.
  Score range: minimum 2.0, maximum 36.0. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- "Filippo Del Ponte" Hospital, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided